CLINICAL TRIAL: NCT06375512
Title: A Phase 1, Randomized, Multicenter, Double-blind, Dose-ranging Study to Evaluate the Safety, Reactogenicity, and Immunogenicity of Herpes Zoster IN001 mRNA Vaccine (IN001) in Healthy Participants 50 to 69 Years Old
Brief Title: A Study to Describe the Safety, Reactogenicity, and Immunogenicity of Herpes Zoster IN001 mRNA Vaccine (IN001) in Healthy Participants
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shenzhen Shenxin Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IN001001
Record Dates: First submitted 2024-04-17; First posted 2024-04-19 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Herpes Zoster
Keywords: IN001; mRNA Vaccine; Vaccine; Varicella-zoster Virus; VZV; Viral Diseases; Shingles; Messenger RNA; Herpes Zoster (HZ); Skin Diseases, Infectious; Safety; Reactogenicity; Immunogenicity; Innorna; Shenxin; Herpesviridae Infections; DNA Virus Infections; Infections; Varicella Zoster Virus Infection; Skin Diseases, Viral; Skin Diseases
MeSH Terms: conditions — Herpes Zoster; Chickenpox; Virus Diseases; Skin Diseases, Infectious; Herpesviridae Infections; DNA Virus Infections; Infections; Varicella Zoster Virus Infection; Skin Diseases, Viral; Skin Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Arm 1: Dose A (Experimental): Participants will receive placebo by intramuscular (IM) injection on Day 0 followed with IN001 by IM injection on Day 56.
  Interventions: Biological: HZ Vaccine (IN001); Biological: Placebo
- Arm 2: Dose B (Experimental): Participants will receive IN001 by IM injection on Day 0 and Day 56.
  Interventions: Biological: HZ Vaccine (IN001)
- Arm 3: Dose C (Experimental): Participants will receive IN001 by IM injection on Day 0 and Day 56.
  Interventions: Biological: HZ Vaccine (IN001)
- Arm 4: Dose D (Experimental): Participants will receive IN001 by IM injection on Day 0 and Day 56.
  Interventions: Biological: HZ Vaccine (IN001)
- Arm 5: Shingrix (Active Comparator): Participants will receive Shingrix by IM injection on Day 0 and Day 56.
  Interventions: Biological: Shingrix

INTERVENTIONS:
Biological: HZ Vaccine (IN001) — Formulation for injection
  Arms: Arm 1: Dose A; Arm 2: Dose B; Arm 3: Dose C; Arm 4: Dose D
Biological: Placebo — 0.9% sodium chloride (normal saline) for injection
  Arms: Arm 1: Dose A
Biological: Shingrix — Sterile suspension for injection
  Arms: Arm 5: Shingrix

SUMMARY:
The study will evaluate the safety, tolerability, and immunogenicity (your immune system's reaction) of the study vaccine called Herpes Zoster IN001 mRNA Vaccine (IN001) in healthy participants who are between 50 and 69 years of age

ELIGIBILITY:
Key Inclusion Criteria:

1. Healthy male or female participants aged between 50 to 69 years of age, inclusive.
2. Body weight ≥ 50 kg for males and ≥ 45 kg for females and body mass index (BMI) in the range of 18.5 to 35 kg/m^2.
3. Participants with asymptomatic medical conditions (eg, hypertension, dyslipidemia) that are not associated with end-organ damage may be included provided they are being appropriately treated as per standard of care, are clinically stable, and are not receiving treatments that would be exclusionary in the opinion of the Investigator.
4. For all women of childbearing potential (WOCBP) females must be non-pregnant and non-lactating and must use a highly effective contraceptive method from at least 30 days prior to enrollment through to 6 months after second vaccination.
5. Willing to provide documented informed consent and comply with the requirements of the clinical study protocol.

Key Exclusion Criteria:

1. Participants with a known history of HZ.
2. Participants with a known history of GBS, encephalomyelitis, or transverse myelitis.
3. Participants with a known history of heart disease (eg, heart failure, recent coronary artery disease, myocarditis, pericarditis, or cardiomyopathy).
4. Participants with acute medical illness or febrile illness, including oral temperature ≥ 38.0°C (≥ 100.4°F) within 1 day prior to screening. Participants with suspected or confirmed COVID-19 should be excluded and referred for medical care.
5. Participants with any medical, neurological, or psychiatric condition that, in the opinion of the Investigator, could place the participant at an unacceptable risk of injury or render the participant unable to comply with all study procedures and achieve successful completion of the trial.
6. Participants with a known history of hypersensitivity reactions including anaphylaxis and urticaria, or other significant adverse reactions to IN001 or its excipients; or participants with a known history of severe allergic reaction (eg, anaphylaxis) to any component of SHINGRIX™ or after a previous dose of SHINGRIX™.
7. Participants who have a positive pregnancy test at the screening visit or who intend to become pregnant during or breastfeed through Study Day 236 (6 months after second vaccination).
8. Participants with uncontrolled hypertension (supine systolic blood pressure ≥ 140 mmHg or supine average diastolic blood pressure ≥ 90 mmHg at screening).
9. Participants with a history of significant hematologic abnormalities or history of thrombosis with thrombocytopenia syndrome.
10. Participants with hematology and/or clinical chemistry laboratory result(s) that meet the definition of a Grade ≥ 2 abnormality as delineated in the FDA guidance.
11. Participants with a history of congenital or acquired immunodeficiency.
12. Participants with an immunosuppressive or immunodeficient state, asplenia, or recurrent severe infections.
13. Participants with a known history of chronic infection including, but not limited to, human immunodeficiency virus (HIV), hepatitis B virus (HBV), hepatitis C virus (HCV), and active tuberculosis.
14. Positive HBV and HCV panel and/or positive HIV test.
15. Participants with positive syphilis test.
16. Participants with chronic illness that, in the opinion of the Investigator, is at a stage where it might interfere with trial participation or interpretation of study results.
17. Participants with a known history of vaccination against varicella or HZ.
18. Participants who have received immunoglobulins and/or any blood or blood products within 4 months before the first study vaccination or who plan to receive such products at any time during the study.
19. Participants who have received immunomodulatory, immunostimulatory, or immunosuppressant drugs including interferon and cytotoxic drugs within 3 months of screening (or 5 half-lives, whichever is longer) or who plan to receive them across the duration of the study.
20. Participants requiring systemic corticosteroids exceeding 10 mg/day of prednisone equivalent for ≥ 10 days within 30 days of screening. The use of topical, ophthalmic, inhaled, and intranasal steroid preparations will be permitted.
21. Participants who have received or plan to receive any licensed vaccine ≤ 28 days prior to the first vaccination (Day 0) or who plan to receive a licensed vaccine ≤ 28 days after the first study vaccination or ≤ 28 days before or after the second study vaccination. The only exception is licensed inactivated influenza vaccine or non-replicating influenza vaccine, which may be given ≥ 14 days before or ≥ 28 days after receipt the first or second study vaccination.
22. Participants receiving treatment with another investigational drug, biological agent, or device ≤ 28 days of screening, or 5 half-lives of the investigational drug, whichever is longer; or currently enrolled in or plans to participate in another clinical trial with an investigational agent during the study period (including the follow-up period of the study).
23. Participants with history of drug abuse within 1 year prior to screening or recreational use of soft drugs (such as marijuana) within 1 month or hard drugs (such as cocaine, phencyclidine, opioid derivatives including heroin, and amphetamine derivatives) within 3 months prior to screening.
24. History of alcohol abuse within 1 year prior to screening or regular use of alcohol within 6 months prior to screening that exceeds 10 units for women or 15 units for men of alcohol per week.
25. Positive alcohol breath test result or positive urine drug screen at screening and Study Day 0.
26. Participants who are Investigator site staff members, employees of the Sponsor or the clinical research organization directly involved in the conduct of the study, or site staff members otherwise supervised by the Investigator or immediate family members of any of the previously mentioned individuals.
27. Participants with a demonstrated inability to comply with the study procedures.

Ages: 50 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-07-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Reporting Solicited Local Reactions | For 14 days after each vaccination
Percentage of Participants Reporting Solicited Systemic Reactions | For 14 days after each vaccination
Percentage of Participants With Unsolicited Adverse Events (AEs) | For 28 days after each vaccination
Percentage of Participants With Any Medically Attended AEs (MAAEs) | From initial vaccination to 6 months after the second vaccination
Percentage of Participants With Any Serious Adverse Events (SAEs), Adverse Events of Special Interest (AESIs), AEs Leading to Vaccine Discontinuation, and AEs Leading to Study Withdrawal | From initial vaccination to 12 months after the second vaccination

SECONDARY OUTCOMES:
Geometric Mean Concentration (GMC) of Anti-glycoprotein E (gE) Antibodies as Measured by Enzyme-Linked Immunosorbent Assay (ELISA) | Baseline (before first vaccination); 28 and 56 days post-first vaccination; 14 and 28 days and 3, 6 and 12 months post-second vaccination
Change from Baseline in Geometric Mean Fold Rise (GMFR) of Anti-gE Antibodies as Measured by ELISA | 28 and 56 days post-first vaccination; 14 and 28 days and 3, 6 and 12 months post-second vaccination
Proportion of Participants with Vaccine Response in Anti-gE Antibodies as Measured by ELISA | 28 and 56 days post-first vaccination; 14 and 28 days and 3, 6 and 12 months post-second vaccination
Geometric Mean Titer (GMT) of Anti-VZV Neutralizing Antibodies as Measured by Neutralization Assay | baseline (before first vaccination); 56 days post-first vaccination; 28 days and 6 and 12 months post-second vaccination
Change from Baseline in GMFR of Anti-VZV Neutralizing Antibodies as Measured by Neutralization Assay | 56 days post-first vaccination; 28 days and 6 and 12 months post-second vaccination
Proportion of Participants with Vaccine Response in Anti-VZV Neutralizing Antibodies as Measured by Neutralization Assay | 56 days post-first vaccination; 28 days and 6 and 12 months post-second vaccination
gE-specific T Cell Response (IFN-γ and IL-4 Secreting T Cells) as Measured by Enzyme-Linked Immunospot (ELISpot) | Baseline (before first vaccination); 28 and 56 days post-first vaccination; 28 days and 3, 6 and 12 months post-second vaccination
Frequencies of gE-specific CD4+ and CD8+ T Cells Expressing Activation Markers (i.e., IFN-γ, IL-2, TNFα, CD40L) as Measured by Intracellular Cytokine Staining (ICS) | Baseline (before first vaccination); 56 days post-first vaccination; 14 and 28 days post-second vaccination

CONTACTS AND LOCATIONS:
Locations (3):
- CenExel, Hollywood, Florida, United States
- Australia (2):
  - Emeritus Research Pty Ltd, Sydney, New South Wales
  - Emeritus Research Pty Ltd, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: Undecided